CLINICAL TRIAL: NCT03968848
Title: A Phase 1, Open-Label, Single-Dose Study to Investigate the Influence of Severe Hepatic Impairment on the Pharmacokinetics of Acalabrutinib and Its Metabolite (ACP-5862)
Brief Title: Investigate the Influence of Severe Hepatic Impairment on the Pharmacokinetics of Acalabrutinib and Its Metabolite
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Acerta Pharma BV (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACE-HI-102
Record Dates: First submitted 2019-05-15; First posted 2019-05-30 (Actual); Results first posted 2021-09-10 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-07

CONDITIONS: Hepatic Impairment; Hepatic Insufficiency; Healthy Subjects
Keywords: Hepatic; Acalabrutinib
MeSH Terms: conditions — Hepatic Insufficiency | interventions — acalabrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Subjects with Severe Hepatic Impairment (Experimental): Subjects with severe hepatic impairment (score of 10 to 15 on the Child-Pugh scale) will be administrated a 50-mg single oral dose of acalabrutinib.
  Interventions: Drug: acalabrutinib
- Matched-Control Subjects (Experimental): Subjects with normal hepatic function will be administrated a 50-mg single oral dose of acalabrutinib.
  Interventions: Drug: acalabrutinib

INTERVENTIONS:
Drug: acalabrutinib — A 50-mg single oral dose of acalabrutinib will be administered.

SUMMARY:
This study is investigate the influence of severe hepatic impairment on the pharmacokinetics of acalabrutinib and its metabolite.

ELIGIBILITY:
Inclusion Criteria

* Women must be of non childbearing status
* Understands the study procedures in the ICF and be willing and able to comply with the protocol.
* Willingness and ability to swallow study drug capsule.
* Adult men or women, 18 to 75 years of age

Hepatic-Impaired Subjects Only:

* Subject has a diagnosis of chronic, stable HI.
* Subject's score on the Child-Pugh scale must range from 10 to 15 at screening.

Exclusion Criteria

* History or presence of clinically significant or unstable medical or psychiatric condition or disease in the opinion of the PI.
* Dosed in another clinical trial within 28 days before dosing of study drug and throughout the current study.
* History or presence of drug abuse within 2 years before screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-11-12 (Actual); Primary Completion 2019-03-13 (Actual); Study Completion 2019-03-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Research Site, Miami, Florida
  - Research Site, Orlando, Florida
  - Research Site, Knoxville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=ACE-HI-102&attachmentIdentifier=8655882d-974a-4d05-b3ae-39c27691e65e&fileName=ACE-HI-102_Final_SAP_25Apr2019_REDACTED.pdf&versionIdentifier=
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=ACE-HI-102&attachmentIdentifier=2213f411-0d84-4ee1-8ae4-4b7c9c46a5d4&fileName=ACE-HI-102_Final_Protocol_04Jun2018_RED_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Groups:
- Severe Hepatic Impairment: Subjects with severe hepatic impairment receiving a single dose of 50 mg acalabrutinib (1 x 50 mg capsules)
- Normal Hepatic Function: Subjects with normal hepatic function receiving a single dose of 50 mg acalabrutinib (1 x 50 mg capsules)
Period: Overall Study
Arm/Group | Severe Hepatic Impairment | Normal Hepatic Function
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Severe Hepatic Impairment | Normal Hepatic Function | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.6 (7.96) | 57.1 (4.88) | 57.4 (6.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 7 | 7 | 14
Race/Ethnicity, Customized [Number; unit: Participants]
  Not Hispanic or Latino | 4 | 5 | 9
  Hispanic or Latino | 4 | 3 | 7
Race/Ethnicity, Customized [Number; unit: Participants]
  Black or African American | 0 | 1 | 1
  White | 8 | 7 | 15
Region of Enrollment [Number; unit: Participants]
  USA | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Plasma Acalabrutinib PK Parameters
Description: Area Under the Concentration-Time Curve
Time Frame: Severe HI: pre-dose, and 0.167, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 14, 24, 36, 48, 60, 72 hrs post-dose. Normal HI: pre-dose, and 0.167, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 14, 24 hrs post-dose.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Severe Hepatic Impairment | Normal Hepatic Function
Number analyzed (Participants) | 8 | 8
ng*hr/mL
  AUC0-24 | 1167 (53.6) | 226.1 (55.3)
  AUC0-last | 1161 (53.9) | 220.0 (57.3)
  AUC0-inf | 1169 (53.8) | 226.5 (55.1)

2. Primary Outcome: Maximum Plasma Acalabrutinib Concentration
Description: Maximum Cmax
Time Frame: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Severe Hepatic Impairment | Normal Hepatic Function
Number analyzed (Participants) | 8 | 8
ng/mL | 726.0 (56.2) | 147.7 (116.8)

ADVERSE EVENTS:
Time Frame: From first dose of study drug until 30 days post last dose
Arm/Group | Severe Hepatic Impairment | Normal Hepatic Function
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 1/8 | 0/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Severe Hepatic Impairment (N=8) | Normal Hepatic Function (N=8)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-06-04): https://cdn.clinicaltrials.gov/large-docs/48/NCT03968848/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-25): https://cdn.clinicaltrials.gov/large-docs/48/NCT03968848/SAP_001.pdf